CLINICAL TRIAL: NCT03658343
Title: An Exploratory, Pilot Study Evaluating T2* Imaging for Adult Sarcoma
Brief Title: T2* MRI Analysis for Sarcoma
Status: Completed | Type: Observational
Sponsor: Bryan Allen (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Bryan Allen, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201807711; 5P30CA086862 (NIH)
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Radiotherapy; Magnetic Resonance Imaging; Sarcoma
Keywords: soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Magnetic Resonance Imaging; Magnetic Resonance Myelography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue if further surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- T2* Imaging: Participants undergo T2* MRI imaging before beginning their course of radiation therapy and then after completing radiation therapy, about 2 weeks before their surgery.
  Interventions: Diagnostic Test: T2* Imaging

INTERVENTIONS:
Diagnostic Test: T2* Imaging — T2* imaging sequences for MRI
  Other Names: magnetic resonance imaging; T2-star; T2* MRI

SUMMARY:
T2* imaging is a method to identify labile iron pools in tumor cells. These iron pools may be linked to better treatment outcomes for specific types of therapy. This is a small pilot study to see if radiation therapy changes the amount of iron in a sarcoma tumor.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed Sarcoma, by biopsy or excision
* prescribed radiation therapy as per standard of care
* treatment to begin within 5 weeks after surgery or biopsy
* ECOG 0, 1, or 2
* ability and willingness to provide informed consent

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically confirmed sarcoma that have been recommended for standard of care radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Change in ferric iron levels detected by T2* MRI | baseline and 8 weeks
  Change from baseline in Fe3+ iron levels

SECONDARY OUTCOMES:
Change in ferrous iron levels detected by T2* MRI | Baseline and 8 weeks
  Change from baseline in Fe2+ iron levels

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Allen, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants may opt in for individual data sharing; the data of those participants who have opted-in will be shared per plan.
Supporting Information: ICF
Time Frame: After completion and analysis of data
Access Criteria: Interested investigators should contact the study PI. Depending upon the data requested, an IRB application may be necessary.